CLINICAL TRIAL: NCT04604262
Title: A Randomised Controlled Clinical Trial to Determine if the Use of the Waterpik in Addition to the Manual Toothbrush Maintains Cleaner Teeth in Patients With Fixed Braces
Brief Title: Does Use of the Waterpik Maintain Cleaner Teeth in Patients With Fixed Braces
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties (due to Covid), no difference found between study arms
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 266235
Record Dates: First submitted 2020-10-09; First posted 2020-10-27 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Intervention Model Description: This will be a 56-week single blind, stratified; parallel group randomised controlled clinical trial. This will be a pseudo-longitudinal trial where observations are recorded at certain fixed intervals.
Who Masked: Outcomes Assessor
Masking Description: Independent outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Waterpik® in addition to the manual toothbrush
  Interventions: Device: Waterpik
- Control (No Intervention): Manual toothbrush

INTERVENTIONS:
Device: Waterpik — Waterpik dental water jet
  Arms: Treatment Group

SUMMARY:
There is no long term evidence to show that the use of Waterpik® is effective for orthodontic patients with fixed braces. A Cochrane Systematic Review confirms this. The aims of this study is to find out if the use of Waterpik® in addition to the manual toothbrush is better to maintain clean teeth in patients with fixed braces. The null hypothesis is that there is no difference between patients using either Waterpik® in addition to the manual toothbrush (treatment group) when compared with patients using just the manual toothbrush (control group).

DETAILED DESCRIPTION:
This will be a 56-week single blind, stratified; parallel group randomised controlled clinical trial. This will be a pseudo-longitudinal trial where observations are recorded at certain fixed intervals. The CONSORT guidelines for reporting randomised control trials will be followed. Examinations will be conducted at baseline, 8, 32 and 56 weeks with 56 weeks classified as the completion of treatment.

These are patients undergoing active orthodontic treatment involving full upper and lower arch fixed appliance therapy. As the selection criteria are quite complicated, a checklist will be used to ensure conformity.

Selection criteria:

1. All patients will have a dental history that included brushing at least twice a day and be willing and able to comply with the trial regime. They will also be between 10 and 20 years of age and in good general health. Any patients with medical conditions and those necessitating chemotherapy which may alter the oral tissue's response to fixed appliance treatment will be excluded. Examples include heart conditions requiring antibiotic cover, diabetes mellitus, immunosuppressant drugs, antibiotics, steroids and hormonal therapy.
2. Patients with decreased manual dexterity either due to mental or physical disabilities and poor compliance will be excluded. Patients with poor initial periodontal health will also be excluded.
3. All medications which may alter plaque accumulation should be avoided during the trial period, but if required on professional advice should report this to the clinical investigator.
4. All patients will have brackets as opposed to bands except permanent molar teeth which may be banded.
5. The patients will have full upper and lower arch treatment as oppose to sectional arch treatment. This is so that the difficulties involved in cleaning all the teeth are similar.
6. They should be bonded using one single type of cement, as we are unsure if different types of cement would influence the accumulation of plaque. This may be true with glass ionomer cement, as it has been shown to inhibit growth of some bacteria. The cement chosen for this purpose is Transbond XT® by 3M Unitek as this the cement most familiar to the operator. Furthermore any breakages from the appliances will be repaired using this cement. This will also ensure that consistent cement will be used.
7. The fixed braces will be of the pre-adjusted Edgewise type as auxiliaries used in other appliance type may pose to be confounding factor. As this unit uses the AO Orthodontics, MBT prescription brackets, this will be the brackets used for this trial.
8. Patients who already use any other supplements to the manual toothbrush for their oral hygiene will be excluded so as not to disadvantage their oral hygiene during their trial

The gold standard The Gold Standard for orthodontic patients is the use of manual toothbrushes to clean in the inter-bracket areas of the fixed braces after each meal or snack. However, for practical purposes, it may not be possible to do so. Some schools do not provide facilities for their pupils to clean their teeth except for the sinks in the toilet. Therefore, patients will be asked to clean their teeth after breakfast, tea and last thing at night. They will be asked to do so for two minutes each time. They will be asked to time themselves and to keep a diary. They will not be given a timer as this is not in keeping with a "real world" situation.

They will also be shown how to clean around the orthodontic brackets using a manual toothbrush by the dental nurse/hygienist using a model. To ensure conformity, this advice will be given by the same two/three dental nurse on each occasion. The dental nurse would be a qualified dental health educator and would be familiar with providing oral hygiene instruction to patients with fixed appliance therapy. However, no further oral hygiene instructions will be given throughout the duration of the trial.

Additionally, if they live in a non-fluoridated area, a 10 mls 2% Fluoride mouthwash would be advised. They would be advised to do this last thing at night by holding the mouthwash for one full minute and spitting out. They would be asked not to rinse thereafter and to go to bed. Since the North Yorkshire area is non-fluoridated, this advice would follow.

Each subject should be issued with a standard fluoride containing toothpaste, a manual toothbrush and those requiring, a Waterpik®. At each visit, they will be issued with replacement brushes or as recommended by the toothbrush manufacturers. As part of the agreement for the patient to take part, they will be given the fluoride mouth rinse to be used last thing at night. The use of any other oral hygiene implements will not be permitted throughout the duration of the trial. No other members of the family will be allowed to use the implements supplied for the purposes of this trial.

All subjects will be issued with a diary of their cleansing habits to encourage motivation and compliance. Only patients who showed good compliance at the preliminary discussion and instruction will be allowed to participate in the trial.

All the instructions will be reinforced by a printed handout.

ELIGIBILITY:
1. All patients will have a dental history that included brushing at least twice a day and be willing and able to comply with the trial regime. They will also be between 10 and 20 years of age and in good general health. Any patients with medical conditions and those necessitating chemotherapy which may alter the oral tissue's response to fixed appliance treatment will be excluded. Examples include heart conditions requiring antibiotic cover, diabetes mellitus, immunosuppressant drugs, antibiotics, steroids and hormonal therapy.
2. Patients with decreased manual dexterity either due to mental or physical disabilities and poor compliance will be excluded. Patients with poor initial periodontal health will also be excluded.
3. All medications which may alter plaque accumulation should be avoided during the trial period, but if required on professional advice should report this to the clinical investigator.
4. All patients will have brackets as opposed to bands except permanent molar teeth which may be banded.
5. The patients will have full upper and lower arch treatment as oppose to sectional arch treatment. This is so that the difficulties involved in cleaning all the teeth are similar.
6. They should be bonded using one single type of cement, as we are unsure if different types of cement would influence the accumulation of plaque. This may be true with glass ionomer cement, as it has been shown to inhibit growth of some bacteria. The cement chosen for this purpose is Transbond XT® by 3M Unitek as this the cement most familiar to the operator. Furthermore any breakages from the appliances will be repaired using this cement. This will also ensure that consistent cement will be used.
7. The fixed braces will be of the pre-adjusted Edgewise type as auxiliaries used in other appliance type may pose to be confounding factor. As this unit uses the AO Orthodontics, MBT prescription brackets, this will be the brackets used for this trial.
8. Patients who already use any other supplements to the manual toothbrush for their oral hygiene will be excluded so as not to disadvantage their oral hygiene during their trial

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Change in Plaque index from baseline | 8, 32, 56 weeks
  The patient will be disclosed by the clinical investigator who will be blind to the toothbrush group allocation. The disclosed mouth will be photographed and plaque scored at the same time. The photograph will allow for a re-score and to check the validity of the clinical score.
  Plaque will be assessed on the buccal surfaces of the teeth on which orthodontic brackets has been placed using the orthodontic modification of the Silness and Loe plaque index. This index has been shown to be sensitive in detecting differences in plaque levels in orthodontic patients with fixed braces. This index divides the tooth surface into four zones in relation to the orthodontic bracket: incisal, distal, mesial and cervical and codes 0-3 were assigned.
Change in Gingivitis from baseline | 8, 32, 56 weeks
  Gingivitis will be measured on the buccal surfaces of the teeth with the gingival index using a CPITN probe.
Change in Gingival bleeding from baseline | 8, 32, 56 weeks
  Gingival bleeding will be determined using the Eastman interdental bleeding index. This will involve inserting a wooden interdental cleaner (Interdental woodsticks, Oral-B Laboratories, Aylesbury, UK) between the teeth from the buccal aspect and depressing the interdental papilla by 1-2 mm. The presence or absence of marginal interdental bleeding from the papilla within 15 seconds will be recorded. The Eastman interdental bleeding index is the number of bleeding sites as expressed as a percentage of the total sites evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- York Teaching Hospital NHS Foundation Trust, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided